CLINICAL TRIAL: NCT06604676
Title: Patient and Operator Centered Outcomes in Harvesting Technique of Soft Tissue Graft: Guided Versus Non-Guided
Brief Title: Patient and Operator Centered Outcomes Concerning Connective Tissue Graft Should Be Considered to Choose Adequately Which Protocol to Use
Acronym: RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, safinaz saleh mohamed saeed, lecturer of periodontics, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #R-OMPDR-2-24-3096
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- guided soft tissue grafting technique (Active Comparator): aguide was fabricated for harvesting the graft and patient and operater centered outcomes is recorded
  Interventions: Procedure: guided soft tissue grafting
- non-guided soft tissue grafting technique (Active Comparator): the graft was taken with the scalpel without guide
  Interventions: Procedure: non-guided soft tissue grafting technique

INTERVENTIONS:
Procedure: guided soft tissue grafting — guided soft tissue grafting techniquea special digital guide was fabricated for one intervention non-guided soft tissue grafting technique receive the traditional technique without guide
  Arms: guided soft tissue grafting technique
Procedure: non-guided soft tissue grafting technique — the graft was taken with traditional technique without guide
  Arms: non-guided soft tissue grafting technique

SUMMARY:
The goal of this clinical trial is to evaluate patient and operator centered outcomes after connective tissue graft harvesting with a fully digital workflow and compare this approach with a conventional one. The main questions it aims to answer are:

* Does it differ in patient- and operator-centered outcomes between the conventional and digital workflow?
* What is the difference in time efficiency between conventional and digital protocols? Researchers will compare digital guided versus conventional technique to choose adequately which protocol to use.

Participants will:

* Receive periodontal surgery to treat gingival recession site
* Visit the clinic after 2 weeks for suture removal & filling the survey
* The time will be recorded during the surgery

DETAILED DESCRIPTION:
50 sites will be included. All investigations will be carried out in accordance with the 1975 Helsinki Declaration, as revised in 2013 for ethical approval. All participants will provide written informed consent after receiving explanations on study objectives and procedures. Primary outcomes will be patient- and operator-centered outcomes. Patient- and operator-centered outcomes will be assessed through visual analogue scale (VAS), questionnaires containing self-developed questions about each phase of the treatment which will be administered at the end of each phase. The questionnaires will be administered as part of a survey which aimed to obtain information about the dental practices. Secondary outcomes will be time-efficiency by assessing workflow duration and number of appointments needed to complete the procedure. The treatment phases will include digital analysis of landmarks and design, of the guide and surgical phase (free gingival graft harvesting ). Time will be recorded in minutes. All the parameters will be recorded in the clinical chart by the same two operators not involved in the treatment after each phase was completed. The planned duration for the research will be 6 months.

ELIGIBILITY:
Inclusion Criteria:

* area need soft tissue augmentation around teeth either coronal or apical to recession
* must have a general health showing no contraindications for oral surgery must be at least 20 years old.
* patients also had to have good oral hygiene before the treatment

Exclusion Criteria:

* signs or symptoms of bruxism or clenching
* if they were suffering from uncontrolled systemic conditions

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Patient- and operator-centered outcomes will be assessed through visual analogue scale (VAS) | 6 months
  Primary outcome will be patient- and operator-centered outcome. Patient- and operator-centered outcome will be assessed through visual analogue scale (VAS).
The questionnaires containing self-developed questions about each phase of the treatment | 6 months
  The questionnaires containing self-developed questions about each phase of the treatment which will be administered at the end of each phase. The questionnaires will be administered as part of a survey which aimed to obtain information about the dental practices.

SECONDARY OUTCOMES:
The time-efficiency by assessing workflow duration | 6 months
  Secondary outcome will be time-efficiency by assessing workflow duration
The number of appointments needed to complete the procedure | 6 months
  Secondary outcome will be number of appointments needed to complete the procedure

CONTACTS AND LOCATIONS:
Overall Officials: bassem nabil elfahl, assistant professor, Principal Investigator — faculty of dentistry,tanta university
Locations (1):
- Faculty of Dentistry ,Tanta University, Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No